CLINICAL TRIAL: NCT04086316
Title: Vulnerable and Resilient Phases During the Menstrual Cycle and Their Influence on Depressive Symptoms and Stress. An Ambulatory Assessment Study on Healthy Women and Women With Depression.
Brief Title: Depressive Symptoms and Subjective Stress in the Course of the Menstrual Cycle - an Ambulatory Assessment Study.
Acronym: DepCy
Status: Completed | Type: Observational
Sponsor: Freie Universität Berlin (Other)
Responsible Party: Principal Investigator, Dr. Sarah Schumacher, Postdoctoral researcher, Freie Universität Berlin
Other Study IDs: CycleDepression
Record Dates: First submitted 2019-08-27; First posted 2019-09-11 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Major Depressive Episode
Keywords: Menstrual Cycle; Major Depressive Disorder; Stress; Sex hormones; Depression; Female; Ambulatory Assessment
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Depression Group: Naturally cycling women with a major depressive episode, assessed by Structured Clinical Interview for DSM-5 (SCID Clinical Version)
- Healthy Group: Naturally cycling women without a major depressive episode, assessed by Structured Clinical Interview for DSM-5 (SCID Clinical Version)

SUMMARY:
Background:

Major changes in female sex hormone concentrations influence the development of depressive symptoms in women. This hypothesis has been thoroughly investigated with regard to the menopause, the postpartal phase and also premenstrual dysphoric disorder. However, much less is known regarding the impact of female sex hormone fluctuations on depression during the regular menstrual cycle. There are indications that during the luteal phase, women might be more vulnerable to the development of depressive symptoms, while during the follicular phase and at ovulation, hormone concentrations might present a protective factor against depressive symptomatology. Subjective stress could mediate the relationship between depressive symptom development and the menstrual cycle phases. The complex interaction between sex hormones and psychological symptoms in the course of menstrual cycle phases is still understudied.

Method:

74 women (37 with and 37 without current depressive episode), will take part in a smartphone-based ambulatory assessment. Women will provide daily ratings of depressive symptoms and perceived stress for a period of one menstrual cycle (approx. 26-30 days). Three menstrual cycle phases will be assessed - the follicular phase, ovulation and the luteal phase. An ambulatory assessment will be used for these daily assessments. To assess the menstrual cycle phase participants will use ovulation tests on five days in the late follicular phase.

The following research questions will be investigated:

Research question 1: Do depressive symptoms (number and severity) change in the course of the menstrual cycle within the two groups? Research question 2: Which depressive symptoms are particularly sensitive to changes in the course of the menstrual cycle phases? Research question 3: Does the subjective stress change in the course of the menstrual cycle within the two groups? Research question 4: Are there differences between depressive and healthy women in terms of changes in depressive symptoms and subjective stress experience?

Implications:

The aim of the study is to investigate women-specific psychobiological factors influencing depression. Therefore, fluctuations in depressive symptoms and subjective stress experience will be investigated as a function of the respective menstrual cycle phases. The identification of cycle phases associated with increased or reduced vulnerability to depressive symptoms will support the development of women-specific prevention and treatment programs.

ELIGIBILITY:
For participants with major depressive episode:

Inclusion criteria:

* female sex
* current diagnosis of a major depression episode
* minimum age of 18 years
* regular menstrual cycle.

Exclusion criteria:

* Pregnancy less than one year ago;
* women who are breastfeeding;
* bipolar disorder;
* acute suicidal tendencies;
* schizophrenic disorders (F20-29);
* substance use disorders
* psychotropic drugs in the last six months;
* chronic somatic diseases.

For participants without major depressive episode:

Inclusion criteria:

* female sex;
* minimum age of 18 years;
* regular menstrual cycle.

Exclusion criteria:

* current or lifetime mental disorder;
* pregnancy less than one year ago;
* women who are breastfeeding;
* psychotropic drugs in the last six months;
* chronic somatic diseases.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Sample will be recruited all over Germany.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Changes in Depressive Symptoms between the menstrual cycle phases | Depressive Symptoms will be assessed daily with an ambulatory assessment for the duration of one menstrual cycle (approx. 28 days).
  Depressive Symptoms will be measured with the Patient Health Questionnaire (PHQ-9), which will be adapted for the ambulatory assessment use (e.g. changing "in the last two weeks" to "right now").
Changes in subjective stress (self report) between the menstrual cycle phases | Subjective stress will be assessed daily with an ambulatory assessment for the duration of one menstrual cycle (approx. 28 days).
  Stress Symptoms will be measured with the short Version of the Perceived Stress Scale (PSS-4), which will be adapted for the ambulatory assessment use (e.g. changing "in the last two weeks" to "right now").

SECONDARY OUTCOMES:
Differences between women with and without a Major depressive Episode | Depressive Symptoms will be assessed daily with an ambulatory assessment for the duration of one menstrual cycle (approx. 28 days).
  Differences between women with and without a Major depressive Episode (measured with the SCID-CV)
Differences between women with and without a Major depressive Episode | Subjective stress will be assessed daily with an ambulatory assessment for the duration of one menstrual cycle (approx. 28 days).
  Differences between women with and without a Major depressive Episode (measured with the SCID-CV)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Schumacher, PhD, Principal Investigator — Freie Universität Berlin
Locations (1):
- Freie Universität Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Klusmann H, Brose A, Schulze L, Engel S, Laufer S, Bucklein E, Knaevelsrud C, Schumacher S. Menstrual cycle related depressive symptoms and their diurnal fluctuations - an ambulatory assessment study. BMC Womens Health. 2024 Nov 18;24(1):611. doi: 10.1186/s12905-024-03438-9. PMID 39551735